CLINICAL TRIAL: NCT06180525
Title: Radiological Evaluation of 3D Printed Porous Collars in Resection Prostheses Hip and Knee: Pilot Study.
Brief Title: Radiological Evaluation of 3D Printed Porous Collars in Hip and Knee Resection Prostheses: Pilot Study.
Acronym: COLLARS
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: San Filippo Neri General Hospital (Other); Istituto Ortopedico Rizzoli (Other); A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Sponsor
Other Study IDs: RS1793/22(2702)
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Bone Tumor
Keywords: Radiological evaluation; Clinical evaluation
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective part: Patients for whom follow-up data up to at least 1 year after surgery is available at the start of the study.
- Prospective part: Both for patients not yet undergoing treatment intervention, at the start of the study, according to the inclusion criteria, both regarding those in follow-up for whom data are not available according to the time of observation required (1 year), will begin once all necessary authorizations have been obtained administrative requests

SUMMARY:
This study aims to evaluate the osseointegration of 3D printed porous collars in hip and knee resection prostheses, in order to eliminate one of the causes of diaphyseal osteolysis, which often lead to loosening of the implants, and therefore to guarantee a further improvement in fixation of the implants in terms of both primary and secondary stability.

DETAILED DESCRIPTION:
Non-interventional, retro-prospective, non-pharmacological multicenter pilot study.

The objective of the study is the radiological and clinical evaluation of collar osteointegration porous 3D printed in hip and knee resection prostheses.

Aims to enroll patients undergoing resection prosthesis surgery hip and knee with the use of 3D printed porous collars, performed according to normal practice clinic at the institutions participating in the study.

It is structured in a retrospective part which will evaluate the patients for whom follow-up data is available at the time of the start of the study up to at least 1 year after the operation. And a prospective part (both with regard to patients not yet subjected to intervention, at the start of the study, according to the inclusion criteria, both regarding those in follow-up for whom data are not available according to the time of observation required (1 year)) which will begin once all the necessary authorizations have been obtained administrative requests.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years at the time of surgery.
* patients undergoing hip and knee resection prosthesis surgery with the use of collars porous 3D printed.
* date of intervention: starting from the regular entry into use of 3D printed porous collars at the reference center.
* Patients operated on for primary tumor outcomes.
* Patients operated on for infection.
* Patients operated for revisions with severe loss of bone substance.
* Patients capable of giving informed consent and obtaining written informed consent (prospective part/patients in follow-up).

Exclusion Criteria:

* Patients lost to follow-up and/or for whom radiographic and clinical documentation is not available corresponding to the post-operative moment and the clinical follow-up visit (6 months and 1 years).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 30 patients will be enrolled consecutively (of which 10 patients consecutively retrospective).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Radiological evaluation | 6 months and 1 year
  Osseointegration will be assessed by x-ray analysis 6 months and 1 year after surgery

SECONDARY OUTCOMES:
QoL evaluation | 6 months and 1 year
  Patient satisfaction/quality of life will be assessed 6 months and 1 year after surgery validated clinical questionnaire (Oxford score).
  Bone remodeling will be evaluated by x-ray analysis 6 months and 1 year after surgery. Number of adverse events of any nature during follow-up. Highlight any inter-observer variability in the detection of radiological measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy